CLINICAL TRIAL: NCT07405723
Title: Arm Position and Blood Pressure Measurement Accuracy in Pregnancy: A Randomized Controlled Trial
Brief Title: Arm Position and Blood Pressure Measurement Accuracy During Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Axelrod, Obstetrician-Gynecologist, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2177-25-SMC; 2177-25-SMC (Other: Sheba Medical Center IRB)
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy; Blood Pressure Measurement in Pregnancy; Hypertensive Disorder of Pregnancy
Keywords: Blood Pressure Measurement; Pregnancy; Arm Position; Hypertensive Disorders of Pregnancy; Prenatal Care; Blood Pressure Accuracy; Randomized Crossover Trial
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Intervention Model Description: Participants undergo blood pressure measurements with the arm placed in multiple positions in a randomized order during a single clinic visit, allowing each participant to serve as her own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm Supported at Heart Level (Experimental): Blood pressure measurements are obtained with the arm supported at heart level while the participant is seated.
  Interventions: Other: Arm Supported at Heart Level
- Arm Supported on Lap (Experimental): Blood pressure measurements are obtained with the arm supported on the participant's lap while seated.
  Interventions: Other: Arm Supported on Lap
- Arm Unsupported at Side (Experimental): Blood pressure measurements are obtained with the arm unsupported at the participant's side while seated.
  Interventions: Other: Arm Unsupported at Side

INTERVENTIONS:
Other: Arm Supported at Heart Level — Blood pressure measurements are obtained with the arm supported at heart level while the participant is seated.
  Arms: Arm Supported at Heart Level
Other: Arm Supported on Lap — Blood pressure measurements are obtained with the arm supported on the participant's lap while seated.
  Arms: Arm Supported on Lap
Other: Arm Unsupported at Side — Blood pressure measurements are obtained with the arm unsupported at the participant's side while seated.
  Arms: Arm Unsupported at Side

SUMMARY:
Accurate blood pressure measurement is essential during pregnancy, as blood pressure readings guide clinical decisions related to the diagnosis and management of hypertensive disorders of pregnancy. Clinical guidelines recommend measuring blood pressure with the arm supported at heart level; however, in routine practice, blood pressure is often measured with the arm in non-standard positions.

This study aims to evaluate how different arm positions affect blood pressure measurements in pregnant women. Pregnant women attending a high-risk pregnancy clinic will undergo blood pressure measurements with the arm placed in several commonly used positions, including supported at heart level, supported on the lap, and unsupported at the side. Each participant will have multiple measurements taken during a single clinic visit.

The study is designed as a randomized crossover trial, allowing each participant to serve as her own control. Participants will be enrolled in trimester-specific cohorts, and results will be analyzed separately for each trimester of pregnancy. The primary outcome is the difference in systolic and diastolic blood pressure measurements between arm positions.

The findings of this study may help improve the accuracy of blood pressure measurement during pregnancy and inform clinical practice regarding optimal measurement techniques.

DETAILED DESCRIPTION:
Blood pressure measurement is a routine and essential component of prenatal care and plays a central role in the diagnosis and management of hypertensive disorders of pregnancy. International and national guidelines recommend measuring blood pressure with the patient seated, after a period of rest, and with the arm supported at heart level. Despite these recommendations, blood pressure in clinical practice is frequently measured with the arm placed in non-standard positions, which may lead to inaccurate readings and potential misclassification of blood pressure status.

This study is designed to assess the effect of arm position on blood pressure measurements in pregnant women. The study consists of three separate prospective randomized crossover trials, each conducted within a specific trimester of pregnancy (first, second, and third trimesters). Participants are enrolled during routine visits to a high-risk pregnancy clinic and are assigned to a trimester-specific cohort based on gestational age at the time of enrollment.

During a single clinic visit, each participant undergoes multiple blood pressure measurements with the arm positioned in several commonly used positions: supported on a desk at heart level, supported on the lap, and unsupported at the side. To account for natural variability in blood pressure measurements, an additional set of measurements with the arm supported at heart level is obtained. The order of arm positions is randomized for each participant using a computerized randomization system, allowing each participant to serve as her own control.

Blood pressure measurements are performed by trained nursing staff using a clinically approved automated blood pressure device, following a standardized measurement protocol. All measurements are obtained after a resting period and while the participant is seated comfortably.

Participants are recruited independently for each trimester cohort, and analyses are conducted separately by trimester. The primary outcome is the difference in systolic and diastolic blood pressure measurements between arm positions. Secondary analyses evaluate the magnitude and pattern of blood pressure differences across gestational ages and relevant clinical subgroups.

This study involves minimal risk and does not alter standard clinical care. The results are intended to improve understanding of how arm positioning influences blood pressure measurements during pregnancy and to inform best practices for accurate blood pressure assessment in prenatal care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 to 55 years
* Singleton or multiple viable intrauterine pregnancy
* Gestational age corresponding to first, second, or third trimester at the time of enrollment
* Ability to sit upright comfortably for the duration of blood pressure measurements
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Preexisting significant cardiac disease (e.g., arrhythmias, congenital heart disease, severe valvular disease)
* Chronic kidney disease defined as serum creatinine ≥1.5 mg/dL at enrollment
* Significant upper limb or shoulder conditions that may affect arm positioning or blood pressure measurement (e.g., lymphedema, fractures, prior surgery, arteriovenous fistula)
* Neurological or musculoskeletal conditions preventing proper positioning
* Severe preeclampsia, eclampsia, or other acute medical conditions requiring immediate intervention
* Major fetal anomaly
* Intrauterine fetal demise

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Systolic and Diastolic Blood Pressure Between Arm Positions | At the study visit (single study visit on the day 1 of enrollment)
  The within-participant difference in mean systolic and diastolic blood pressure measurements obtained with the arm supported at heart level, supported on the lap, and unsupported at the side. Blood pressure values are calculated as the mean of triplicate measurements for each arm position.

SECONDARY OUTCOMES:
Magnitude of Blood Pressure Differences Between Arm Positions | At the study visit (single study visit on the day 1 of enrollment)
  The absolute difference in mean systolic and diastolic blood pressure measurements between each pair of arm positions (supported at heart level, supported on the lap, unsupported at the side), calculated within each participant.
Variation in Blood Pressure Differences Across Gestational Age | At the study visit (single study visit on the day 1 of enrollment)
  Comparison of within-participant differences in systolic and diastolic blood pressure between arm positions across trimester-specific cohorts of pregnancy.
Effect of Arm Position on Blood Pressure by Chronic Hypertension Status | At the study visit (single study visit on the day 1 of enrollment)
  Comparison of within-participant differences in systolic and diastolic blood pressure between arm positions among participants with and without preexisting chronic hypertension.
Comparison of Systolic Versus Diastolic Blood Pressure Sensitivity to Arm Position | At the study visit (single study visit on the day 1 of enrollment)
  Assessment of differences in the magnitude of arm position-related variation between systolic and diastolic blood pressure measurements within participants.
Blood Pressure Differences by Singleton Versus Multiple Pregnancy | At the study visit (single study visit on the day 1 of enrollment)
  Comparison of within-participant differences in systolic and diastolic blood pressure between arm positions in singleton and multiple pregnancies.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data sharing plans have not yet been determined. Any future data sharing will be subject to institutional policies, ethical approvals, and data protection requirements.

REFERENCES:
- [Background] Liu H, Zhao D, Sabit A, Pathiravasan CH, Ishigami J, Charleston J, Miller ER 3rd, Matsushita K, Appel LJ, Brady TM. Arm Position and Blood Pressure Readings: The ARMS Crossover Randomized Clinical Trial. JAMA Intern Med. 2024 Dec 1;184(12):1436-1442. doi: 10.1001/jamainternmed.2024.5213. PMID 39373998